CLINICAL TRIAL: NCT00881608
Title: An Open-Label, Escalating Dose, Single Center, Cross-over Design, Phase I Study to Evaluate Menses Induction in Women Administered Proellex
Brief Title: Study to Evaluate Menses Induction in Women Administered Proellex
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Repros stopped study for safety and the FDA put the study on hold for safety.
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZP-010
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Amenorrhea
Keywords: Menstruation
MeSH Terms: conditions — Amenorrhea | interventions — telapristone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Initiation-Placebo Cycle-Five (5) placebo capsules will be dispensed to subjects to self-administer for five days starting on cycle day 18.
  Interventions: Drug: Placebo
- 3 mg Proellex (Experimental): First Cycle (3 mg)- Five (5) 3 mg capsules of Proellex will be dispensed to subjects to self-administer for five days starting on cycle day 18.
  Interventions: Drug: Proellex
- 6 mg Proellex (Experimental): Second Cycle (6 mg)-Subjects, who have not experienced menses, will have their dose of Proellex escalated, and be dispensed ten (10) 3 mg capsules of Proellex to self-administer 2, 3 mg capsules each day for five days starting on cycle day 18.
  Interventions: Drug: Proellex
- 12 mg Proellex (Experimental): Third Cycle (12 mg)-Subjects, who have not experienced menses, will have their dose of Proellex escalated, and be dispensed twenty (20) 3 mg capsules of Proellex to self-administer 4, 3 mg capsules for five days starting on cycle day 18.
  Interventions: Drug: Proellex
- 25 mg Proellex (Experimental): Fourth Cycle (25 mg)-Subjects, who have not experienced menses, will be dispensed five (5) 25 mg capsules of Proellex to self-administer for five days starting on cycle day 18.
  Interventions: Drug: Proellex

INTERVENTIONS:
Drug: Placebo — Placebo, 1 capsule daily for five days
  Other Names: Dummy
  Arms: Placebo
Drug: Proellex — Proellex, one 3, 6, 12 or 25 mg capsule daily for five days
  Other Names: Telapristone acetate
  Arms: 12 mg Proellex; 25 mg Proellex; 3 mg Proellex; 6 mg Proellex

SUMMARY:
The purpose of this study is to determine the oral dose level at which the investigative drug, Proellex, is able induce menstruation.

DETAILED DESCRIPTION:
The purpose of this study is to determine the oral dose level at which the investigative drug, Proellex, is able to suppress endogenous progesterone in women. It is believed that giving Proellex in the early/mid-luteal phase of the cycle will suppress the effects of endogenous progesterone triggering the end of the cycle and inducing menstruation as happens naturally

ELIGIBILITY:
Inclusion Criteria:

* Clinical laboratory tests within normal ranges
* A normal menstrual period of 26-30 days
* Desiring not to become pregnant
* Agreeing to use a double barrier method of birth control for the duration of the trial

Exclusion Criteria:

* Post-menopausal status
* Aamenorrhea or dysfunctional uterine bleeding
* Subjects demonstrating any clinically significant medical condition rendering the subjects infertile or marginally fertile
* Subjects with a Body Mass Index (BMI) below 18 or over 39

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre van As, M.D., Ph.D, Study Director — Repros Therapeutics Inc.
Locations (1):
- Advances in Health Inc., Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects Enrolled: All subjects initiated treatment with placebo. Further information is not availasble due to premature termination of the study.
Period: Overall Study
Arm/Group | All Subjects Enrolled
Started | 11
Completed | 0
Not Completed | 11
Not completed — Study prematurely terminated | 11

BASELINE CHARACTERISTICS:
Population: Study prematurely terminated, no data available
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 3 mg Proellex | 6 mg Proellex | 12 mg Proellex | 25 mg Proellex | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
Age, Categorical [Count of Participants; unit: Participants]
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Day of Initial Vaginal Bleeding Event Following Treatment With Proellex.
Time Frame: An early vaginal bleeding event lasting at least two days and occurring on or before day 24 will be deemed to have achieved an induced menses
Population: Study prematurely terminated
Arm/Group | Placebo | 3 mg Proellex | 6 mg Proellex | 12 mg Proellex | 25 mg Proellex
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Duration of Vaginal Bleeding Following Treatment With Proellex.
Time Frame: At least 2 days
Population: Study prematurely terminated
Arm/Group | Placebo | 3 mg Proellex | 6 mg Proellex | 12 mg Proellex | 25 mg Proellex
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: No adverse event data is available.
Arm/Group | Placebo | 3 mg Proellex | 6 mg Proellex | 12 mg Proellex | 25 mg Proellex
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated for safety reasons (Proellex studies were put on clinical hold due to liver toxicity). Sponsor was unable to pay vendor, and was therefore not provided with any study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights